CLINICAL TRIAL: NCT07300800
Title: Evaluating The Efficacy of Platelet Rich Plasma on Voice Outcomes Following Surgical Removal of Benign Vocal Fold Lesions
Brief Title: Effect of PRP Injection on Voice Recovery After Benign Vocal Fold Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Shaimaa A Bakia, Lecturer of Phoniatrics, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMBSUREC/04032025/Mohammed
Record Dates: First submitted 2025-12-04; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Benign Vocal Fold Lesions
Keywords: Vocal fold polyps Vocal fold cysts Vocal fold nodules Vocal fold atrophy Vocal fold sulcus Vocal fold scar

STUDY DESIGN:
Intervention Model Description: The surgery will be performed under general anesthesia. All patients will undergo microlaryngoscopic removal of the vocal fold lesions under microscopic or endoscopic guidance using a rigid laryngoscope, and hemostasis will be achieved. For patients in the PRP group, 1.5 mL of PRP will be injected into the superficial lamina propria (Reinke's space), just lateral to the excision site, using a Chiba needle. This site is chosen to promote tissue regeneration without damaging the vocal ligament or muscle, while slightly medializing the vocal fold for better glottic closure. Care will be taken to avoid the free edge of the vocal fold, as direct injection there can cause scarring, stiffness, or worsening of voice quality. The injection volume will typically range from 0.5 to 1.5 mL depending on the size of the lesion and the vocal fold.
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessors / Voice Analysts: masked to group assignment to avoid assessment bias when evaluating voice outcomes (GRBAS, VFI, acoustic analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Group (Experimental): Patients in this group will undergo microlaryngoscopic removal of benign vocal fold lesions followed by an injection of 1.5 mL of platelet-rich plasma (PRP) into the superficial lamina propria (Reinke's space) just lateral to the excision site. This intervention aims to promote tissue regeneration, improve vocal fold healing, and enhance postoperative voice outcomes.
  Interventions: Procedure: Platelet-Rich Plasma (PRP) Injection after Microlaryngoscopic Surgery for PRP Group
- Conventional Surgery Group (Active Comparator): Control (Conventional Surgery) Group
  Role: Control group for comparison.
  Description: Patients in this group will undergo microlaryngoscopic removal of benign vocal fold lesions without PRP injection. Standard postoperative care will be provided. This arm serves as the baseline to assess the additional effect of PRP on voice recovery and healing.
  Interventions: Procedure: Conventional Microlaryngoscopic Surgery (Active Comparator)

INTERVENTIONS:
Procedure: Platelet-Rich Plasma (PRP) Injection after Microlaryngoscopic Surgery for PRP Group — Platelet-Rich Plasma (PRP) Injection Patients in this group will undergo microlaryngoscopic removal of benign vocal fold lesions under general anesthesia. Following surgery, 1.5 mL of autologous PRP will be injected into the superficial lamina propria (Reinke's space), just lateral to the excision site, using a Chiba needle. The injection aims to promote tissue regeneration, improve postoperative healing, and enhance vocal quality. Care is taken to avoid the free edge of the vocal fold to minimize scarring or stiffness. The PRP is prepared fresh from the patient's blood on the day of injection.
  Arms: PRP Group
Procedure: Conventional Microlaryngoscopic Surgery (Active Comparator) — Patients in this group will undergo microlaryngoscopic removal of benign vocal fold lesions under general anesthesia without PRP injection. Standard postoperative care is provided. This group serves as a comparator to evaluate the additional effect of PRP on voice recovery.
  Arms: Conventional Surgery Group

SUMMARY:
The goal of this clinical trial is to evaluate whether platelet-rich plasma (PRP) injections can improve voice outcomes after microlaryngosurgery in patients with benign vocal fold lesions. The main questions it aims to answer are:

Does postoperative PRP injection improve vocal quality compared to conventional surgery alone?

Does PRP injection reduce vocal fatigue and improve patients' voice-related quality of life?

Researchers will compare 32 patients receiving PRP injections after surgery to 32 patients undergoing conventional surgery without PRP to see if PRP enhances recovery and voice function.

Participants will:

Undergo microlaryngosurgery to remove benign vocal fold lesions.

Receive either a PRP injection to the operated vocal fold or standard postoperative care.

Complete voice assessments before surgery and at 1 and 3 months after surgery, including:

Auditory perceptual evaluation (GRBAS scale) Videostroboscopy Acoustic and aerodynamic voice analysis Vocal Fatigue Index (VFI)

All participants will provide written consent and undergo standard preoperative assessments including medical history, ENT examination, laboratory tests, ECG, and anesthesia evaluation.

DETAILED DESCRIPTION:
Benign vocal fold lesions are commonly treated with microlaryngosurgery when conservative management fails; however, postoperative voice recovery may be variable, and some patients experience persistent dysphonia or vocal fatigue. Platelet-rich plasma (PRP) has been proposed as a biologic adjunct that may enhance tissue healing through its regenerative and anti-inflammatory properties.

This clinical trial evaluates the effect of postoperative PRP injection as an adjunct to microlaryngosurgery for benign vocal fold lesions. The study compares voice recovery in patients receiving PRP injection following surgery with those receiving conventional postoperative management alone.

Adult patients undergoing microlaryngosurgery for benign vocal fold lesions will be enrolled and allocated to one of two study groups: a PRP injection group or a conventional treatment group. All participants will undergo standard surgical management, with the intervention group receiving an additional PRP injection to the operated vocal fold.

Voice outcomes will be assessed longitudinally at predefined postoperative intervals using objective, perceptual, and patient-reported measures. These assessments are intended to evaluate postoperative voice quality, vocal function, and patient-perceived vocal fatigue.

All participants will undergo routine preoperative evaluation and provide written informed consent in accordance with institutional and ethical guidelines.

This study aims to determine whether PRP injection provides additional benefit in voice recovery following microlaryngosurgery for benign vocal fold lesions.

ELIGIBILITY:
* Inclusion Criteria:

  * Adults aged 18 to 50 years

  * Diagnosis of a benign vocal fold lesion, including: Vocal fold polyps Vocal fold cysts Vocal fold nodules Vocal fold atrophy Vocal fold sulcus Vocal fold scar

  * Failure to respond to conservative management, including one or more of the following: Voice rest, voice therapy
* Exclusion Criteria:

  * Age younger than 18 years or above 50
  * Medically unfit for surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Shimmer (Local, dB) | From enrollment, including baseline voice assessment, through surgery and postoperative follow-up assessments at 1 month and 3 months
  Shimmer (local), expressed in decibels (dB), representing cycle-to-cycle amplitude variation, will be obtained from sustained vowel /a/ using PRAAT software.

SECONDARY OUTCOMES:
Mean Noise-to-Harmonics Ratio (NHR) | Baseline (preoperative), 1 month postoperative, and 3 months postoperative
  Mean Noise-to-Harmonics Ratio (NHR), a unitless acoustic measure reflecting the proportion of noise relative to harmonic components in the voice signal, will be obtained from sustained vowel /a/ using PRAAT software.
  Unit of Measure:
  Unitless ratio

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Ahmed Bakia, Principal Investigator — Lecturer of Phoniatrics

IPD SHARING:
Plan to Share IPD: No